CLINICAL TRIAL: NCT01946113
Title: Phosphate, Magnesium and Calcium-Homeostasis in Patients With Acute Renal Failure and Continuous Renal Replacement Therapy
Brief Title: Mineral-Homeostasis in Continuous Renal Replacement Therapy
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Prof. Kindgen-Milles, Heinrich-Heine University, Duesseldorf
Other Study IDs: 4209
Record Dates: First submitted 2013-09-09; First posted 2013-09-19 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospektive Cohort: Patients requiring renal replacement therapy from 2011 to 2012 on intensive care unit
- Prospektive Cohort: Patients requiring renal replacement on intensive care unit in 2013 and 2014

SUMMARY:
Acute renal failure is a common complication in intensive care unit patients. In 10% of cases renal replacement therapy becomes necessary. Current devices have increase filter patency and efficacy. However, magnesium, calcium and phosphate are eliminated as well. However, the extend of this elimination hase not been quantified. Thus, we want to

1. record retrospectively how often abnormal values for phosphate, magnesium and calcium occurred during routine renal replacement therapy in 2011 and 2012.
2. prospectively evaluate the same parameters during routine treatment in 2013 and 2014

ELIGIBILITY:
Inclusion Criteria:

* intensive care unit patients with acute renal failure undergoing continuous renal replacement therapy
* older than 18 years of age

Exclusion Criteria:

* age less than 18 years
* pregnancy
* contraindications against continuous renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care unit patients with acute renal failure undergoing renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of hypo-phosphate,-magnesium and calcaemia | approximately 28 days
  Participants will be followed for the duration of ICU stay, an expected average of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Kindgen-Milles, Prof., Principal Investigator — Department of Anaesthesiology, Duesseldorf University Hospital
Locations (1):
- Interdisziplinäre Intensivstation Universitätsklinikum Düsseldorf, Düsseldorf, Germany